CLINICAL TRIAL: NCT01415128
Title: A PHASE I, SINGLE-CENTER, OPEN-LABEL, CROSSOVER STUDY OF THE EFFECT OF AVANAFIL ON THE PHARMACOKINETICS OF OMEPRAZOLE, DESIPRAMINE AND ROSIGLITAZONE IN HEALTHY MALE SUBJECTS
Brief Title: Compare the Pharmacokinetics of Omeprazole, Rosiglitazone, and Desipramine When Administered With Avanafil in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VIVUS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA-018
Record Dates: First submitted 2010-03-28; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Omeprazole; Rosiglitazone; Desipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omeprazole (Active Comparator): Omeprazole with single dose of avanafil (200 mg)
  Interventions: Drug: Omeprazole
- Rosiglitazone (Active Comparator): Rosiglitazone with single dose of avanafil (200 mg)
  Interventions: Drug: Rosiglitazone
- Desipramine (Active Comparator): Desipramine with single dose of avanafil (200 mg)
  Interventions: Drug: Desipramine

INTERVENTIONS:
Drug: Omeprazole — Once a day dosing of Omeprazole (40 mg) for 8 days
  Arms: Omeprazole
Drug: Rosiglitazone — Single dose of Rosiglitazone (8 mg) for 1 day
  Arms: Rosiglitazone
Drug: Desipramine — Single dose of Desipramine (50 mg) for 1 day
  Arms: Desipramine

SUMMARY:
This study will compare the pharmacokinetics of omeprazole, rosiglitazone and desipramine when administered with a single oral dose of avanafil in healthy male subjects.

DETAILED DESCRIPTION:
There will be three cohorts in this Phase I, single-center, open-label, crossover study:

Cohort A (omeprazole): This is a open-label, non-randomized, one-sequence crossover study design, in which 20 healthy male subjects will be enrolled and administered a single oral dose of 40 mg omeprazole once daily for 8 days (Days 1-8) plus a single oral dose of 200 mg avanafil on Day 8. On Days 7 and 8, avanafil and/or omeprazole doses will be administered following an overnight fast of at least 10 hours.

All subjects will be confined at the Clinical Research Unit the day prior to the omeprazole administration on Day 7 and will remain confined for approximately 13 hours following the dosing on Day 8. Blood samples for determination of plasma omeprazole concentrations will be obtained from all subjects at 0 (10 minutes pre-dose), 20, 40 minutes and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 and 12 hours post-dose on Days 7 and 8. Pre-dose blood samples for determination of omeprazole will also be taken in the morning on Days 5-6.

Cohort B (rosiglitazone): This is a randomized, open-label, two-period crossover study design, in which 20 male subjects will be randomized to receive the following treatments:

* Treatment A: a single oral dose of 8 mg rosiglitazone following an overnight fast of at least 10 hours.
* Treatment B: a single oral dose of 8 mg rosiglitazone plus a single oral dose of 200 mg avanafil following an overnight fast of at least 10 hours.

The two treatments in the cohort will be separated by a washout period of at least 7 days. All subjects will be confined at the Clinical Research Unit approximately from the morning of Day -1 to the morning of Day 2 in both treatment periods. Blood samples for determination of plasma rosiglitazone concentrations will be obtained from all subjects at 0 (10 minutes pre-dose) and 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 16 and 24 hours post-dose.

Cohort C (desipramine): This is a randomized, open-label, two-period, crossover study design, in which 20subjects identified as CYP2D6 extensive metabolizers (determined by genotyping) will be randomized to receive the following treatments:

* Treatment A: a single oral dose of 50 mg desipramine following an overnight fast of at least 10 hours.
* Treatment B: a single oral dose of 50 mg desipramine plus a single oral dose of 200 mg avanafil following an overnight fast of at least 10 hours. The avanafil dose will be administered 2 hours after the desipramine administration.

The two treatments in the cohort will be separated by a washout period of at least 10 days. All subjects will be confined at the Clinical Research Unit from the morning of Day -1 to the morning of Day 2 in both treatment periods. Blood samples for determination of plasma desipramine concentrations will be obtained from all subjects at 0 (10 minutes pre-dose) and 1, 2, 4, 6, 8, 10, 12, 24, 48, 72 and 96 hours post-dose. Subjects will visit the study site as outpatients in the morning for their remaining PK blood sample collection on Days 3-5.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily consent to participate in the study (informed consent form must be signed and dated prior to any study related assessments).
2. Adult male subjects of 18 to 45 years of age inclusive.
3. A body weight of at least 50 kg and a body mass index (BMI) between 18 and 30 kg/m2, inclusive [BMI will be calculated as weight in kg/(height in m)2].
4. Subjects must be identified as CYP2D6 extensive metabolizers (determined by genotyping) for Cohort C only
5. Subjects are able to communicate with the investigator, and to understand and comply with all requirements of study participation.
6. Medically healthy, with no clinically significant screening results (e.g., laboratory profiles, medical histories, ECGs, physical exam, etc.), in the opinion of the investigator in consultation with the Sponsor.
7. Male subjects should be willing to use a condom and spermicide during sexual activity for 90 days after last dosing of avanafil and be willing to not donate sperm for 90 days after dosing.

Exclusion Criteria:

1. A history or presence of significant cardiovascular (including thromboembolic disorders), neurological, hematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs or place the subjects at increased risk as determined by the investigator.
2. Any clinically significant laboratory abnormalities as judged by the investigator. Inclusion of a subject with out of normal range laboratory values must be approved by VIVUS prior to subject enrollment.
3. A predisposition to priapism, such as subjects with sickle cell disease or blood dyscrasias.
4. Known history of cardiovascular or cerebrovascular event, any history of angina.
5. History or ECG evidence of any high-risk arrhythmia or ECG judged by the investigator to be clinically significant.
6. Hypertrophic obstructive or other clinically significant cardiomyopathy, moderate or severe cardiac valvular disease.
7. Subjects whose pulse is lower than 50 bpm at screening or 50 bpm prior to dosing for period 1 only.
8. Acute illness, especially any infection, within 2 weeks of dosing.
9. Systolic blood pressure < 90 or > 140 mmHg; diastolic blood pressure < 60 or > 95 mmHg at screening or on Day -1 (2 rechecks are allowed) for period 1 only.
10. History of retinitis pigmentosa or nonarteritic anterior ischemic optic neuropathy.
11. Hemoglobin < 12.0 g/dL.
12. Subjects with liver function tests > 1.5 ULN
13. Positive urine drug test and/or positive urine alcohol test at screening or on Day -1.
14. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV) at screening.
15. Any history or presence of alcoholism or drug or substance abuse within 18 months or as defined by the investigator.
16. Allergy to or previously significant adverse events with PDE5 inhibitors, omeprzole, rosiglitazone and desipramine or their constituents.
17. Use of any prescription or over-the-counter (OTC) medication, including herbal products, within the 30 days prior to Day 1. Up to 2 g per day of acetaminophen is allowed at the discretion of the Investigator.
18. Use of any drug in Appendix 1 (drugs known to have clinical significance in inhibiting or inducing liver enzymes involved in drug metabolism [CYP P450]) within 30 days prior to Day 1.
19. Blood donation or significant blood loss within 56 days prior to Day 1.
20. Plasma donation within 14 days prior to Day 1.
21. Any use of tobacco or nicotine products within 6 months prior to Day 1.
22. Any subject who received an investigational drug within 30 days or six half-lives, whichever is longer, prior to Day 1.
23. Evidence of any clinically significant medical, psychiatric, social or other condition by history, physical examination or laboratory studies that, in the opinion of the investigator, would contraindicate the administration of study medications, affect compliance, interfere with study evaluations, limit study participation, or confound the interpretation of study results.
24. Involvement in the planning and conduct of the study (applies to both VIVUS or designee staff, or staff at the investigational site).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To measure a composite of pharmacokinetic parameters of Omeprazole, Rosiglitazone and Desipramine. | 0, 20, 40 minutes and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 and 12 hours post dose
  AUC0-t, AUC0-inf, Cmax, tmax, half-life

SECONDARY OUTCOMES:
To assess vital signs before, during and after dosing | In the morning at Screening, Days 1-8 and upon early termination
  heart rate and blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, Study Director — VIVUS LLC